CLINICAL TRIAL: NCT01854619
Title: Photodisinfection for the Treatment of Chronic Rhinosinusitis
Brief Title: Photodynamic Therapy for the Treatment of Chronic Rhinosinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ondine Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBI-1212-1
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Sinusitis
Keywords: chronic rhinosinusitis; sinusitis; photodisinfection; photodynamic therapy; antimicrobial photodynamic therapy; aPDT; PDT; paranasal sinus diseases; respiratory tract infections; respiratory tract diseases
MeSH Terms: conditions — Sinusitis; Paranasal Sinus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — Photochemotherapy; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline irrigation (Active Comparator): Saline irrigation via syringe will be administered using a sinus irrigation catheter under endoscopic control.
  Interventions: Device: Saline irrigation
- Double photodisinfection treatment (Active Comparator): Patients in the double treatment arm will receive a second photodisinfection treatment 4 weeks following the first treatment with regular follow-up visits
  Interventions: Device: Photodisinfection (antimicrobial photodynamic therapy, aPDT)
- Single photodisinfection treatment (Active Comparator): The single-treatment group will receive a single photodisinfection treatment of all involved paranasal sinuses with multiple follow-up visits.
  Interventions: Device: Photodisinfection (antimicrobial photodynamic therapy, aPDT)

INTERVENTIONS:
Device: Photodisinfection (antimicrobial photodynamic therapy, aPDT) — A 0.03% solution of methylene blue is irrigated into the involved paranasal sinus followed by placement of a saline filled balloon with a center light diffusing fiber optic. This is illuminated at 150 mW/cm2 power density for 8 minutes. This is repeated for each involved sinus.
  Other Names: PDT; photodynamic therapy; aPDT; light therapy; Sinuwave
  Arms: Double photodisinfection treatment; Single photodisinfection treatment
Device: Saline irrigation — The active comparator arm will receive saline irrigation via syringe that is administered using a sinus irrigation catheter under endoscopic control.
  Other Names: Endoscopic saline irrigation
  Arms: Saline irrigation

SUMMARY:
The purpose of this study is to determine whether the use of light and a topically applied photosensitizer can relieve symptoms and clinically improve patients with chronic rhinosinusitis.

DETAILED DESCRIPTION:
This clinical trial will be a prospective, randomized, single-center study utilizing two treatment assignments and a control group. The study is expected to enroll a total of 48 subjects. The intent of the study is to evaluate a single versus double treatment of photodisinfection in men and women suffering from chronic persistent rhinosinusitis with and without nasal polyposis. Each photodisinfection treatment group will be compared to a control group receiving saline irrigation.

ELIGIBILITY:
Inclusion Criteria:

* history of chronic rhinosinusitis with and without nasal polyposis
* no antibiotics within 4 weeks
* no oral steroid use within 4 weeks
* no topical steroid use within 2 weeks
* endoscopic sinus surgery greater than 6 months previously

Exclusion Criteria:

* acute respiratory infection within last 2 weeks
* septal deviation restricting sinus access
* known allergy to methylene blue
* pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 | 6 months
  The Sino-Nasal Outcome Test (SNOT-22) has been widely adopted in clinical practice and has been proved to be the most suitable and validated sinonasal outcome scoring system. The SNOT-22 is a disease-specific, quality-of-life-related measure of sinonasal function. Low score indicates good outcome.

SECONDARY OUTCOMES:
Microbiome evaluation | 6 months
  Microbiological conventional cultures, gene expression profiling and microbiome profiling by 16s RNA.

OTHER OUTCOMES:
Nasal and sinus symptom score | 6 months
  This is a 5 item subjective list rated by patients from zero to severe.
Endoscopic Evaluation Scoring | 6 months
  This is an endoscopic staging system for non-neoplastic sinonasal disease to evaluate therapeutic outcomes that is complex enough to incorporate the most important measures of the sinonasal cavity but simple enough to facilitate regular clinical use.
CT Scoring | 4 weeks
  The American Academy of Otolaryngology & Task Force on Rhinosinusitis has recommended the Lund-Mackay system as the preferred method of staging of chronic rhinosinusitis (CRS). The Lund-Mackay staging system represents the most widely established method of sinus CT scoring in clinical trials. It scores each sinus area as a 0, 1, or 2 depending on the extent of mucosal opacification present and also includes a score for patency of the ostiomeatal unit.
Smell Testing (UPSIT) | 4 weeks
  The University of Pennsylvania Smell Identification Test (UPSIT) is a scratch and sniff test used in North America since 1984 (Doty, 1984) and is the most widely used olfactory test in the world. The UPSIT is a multiple-forced-choice odour identification test. For each odorant there are four alternative responses and the subject is required to choose one of these even if no smell is perceived. It requires 10-15 min to be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Desrosiers, MD, Principal Investigator — Université de Montréal
Locations (1):
- Centre hospitalier de l'UdeM (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Background] Biel MA, Sievert C, Usacheva M, Teichert M, Balcom J. Antimicrobial photodynamic therapy treatment of chronic recurrent sinusitis biofilms. Int Forum Allergy Rhinol. 2011 Sep-Oct;1(5):329-34. doi: 10.1002/alr.20089. Epub 2011 Aug 18. PMID 22287461
- [Background] Biel MA, Jones JW, Pedigo L, Gibbs A, Loebel N. The effect of antimicrobial photodynamic therapy on human ciliated respiratory mucosa. Laryngoscope. 2012 Dec;122(12):2628-31. doi: 10.1002/lary.23502. Epub 2012 Oct 15. PMID 23070780
- [Background] Biel MA, Pedigo L, Gibbs A, Loebel N. Photodynamic therapy of antibiotic-resistant biofilms in a maxillary sinus model. Int Forum Allergy Rhinol. 2013 Jun;3(6):468-73. doi: 10.1002/alr.21134. Epub 2013 Jan 10. PMID 23307793
- [Background] Krespi YP, Kizhner V. Phototherapy for chronic rhinosinusitis. Lasers Surg Med. 2011 Mar;43(3):187-91. doi: 10.1002/lsm.21042. Epub 2011 Feb 2. PMID 21290392
- [Background] Krespi YP, Kizhner V, Kara CO. Laser-induced microbial reduction in acute bacterial rhinosinusitis. Am J Rhinol Allergy. 2009 Nov-Dec;23(6):e29-32. doi: 10.2500/ajra.2009.23.3404. PMID 19958597